CLINICAL TRIAL: NCT05823766
Title: Transforming Research and Clinical Knowledge in Traumatic Brain Injury Epileptogenesis Project (TRACK-TBI EPI)
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 834420
Record Dates: First submitted 2023-04-10; First posted 2023-04-21 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Traumatic Brain Injury; Post-traumatic Epilepsy
MeSH Terms: conditions — Brain Injuries, Traumatic; Epilepsy, Post-Traumatic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, PAXGene
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Telephone Assessment Battery: TRACK-TBI participants may complete up to three annual telephone calls to assess outcome status and screen for PTE. These assessments will determine eligibility for the in-person study visit.
  Interventions: Behavioral: Telephone Outcome Assessment
- Comprehensive Assessment Battery (CAB): Participants who demonstrate decision-making capacity will be asked to complete the Comprehensive Assessment Battery (CAB). The CAB in-person is comprised of measures of cognition (i.e. attention, memory, information processing speed, executive functions), mood (i.e., depression, anxiety), social participation, subjective well-being, post-traumatic stress, interviews, global functional status measures, and a COVID-19 questionnaire.
  Interventions: Behavioral: In-Person Outcome Assessment; Procedure: 3T Magnetic Resonance Imaging (MRI); Behavioral: Clinical Visit; Procedure: Blood Draw; Procedure: EEG
- Abbreviated Assessment Battery (AAB): Participants who do not have decision-making capacity will be asked to complete a modified assessment battery, called the Abbreviated Assessment Battery (AAB). The AAB in-person assessment will administer the Speech Intelligibility, GOAT, and CAP and/or CRS-R to study participants.
  Interventions: Behavioral: In-Person Outcome Assessment; Procedure: 3T Magnetic Resonance Imaging (MRI); Behavioral: Clinical Visit; Procedure: Blood Draw; Procedure: EEG
- TED Friend Controls: Participants enrolled in the TBI Endpoints Development (TED) cohort from 2017-2019 who did not experience a TBI prior to affiliated enrollment in TRACK-TBI will be asked to complete an assessment battery.
  Interventions: Behavioral: In-Person Outcome Assessment; Procedure: 3T Magnetic Resonance Imaging (MRI); Procedure: Blood Draw

INTERVENTIONS:
Behavioral: In-Person Outcome Assessment — Assessments will be administered to evaluate participant outcome status
  Groups: Abbreviated Assessment Battery (AAB); Comprehensive Assessment Battery (CAB); TED Friend Controls
Procedure: 3T Magnetic Resonance Imaging (MRI) — Participants will be asked to complete a 3T MRI
  Groups: Abbreviated Assessment Battery (AAB); Comprehensive Assessment Battery (CAB); TED Friend Controls
Behavioral: Clinical Visit — Patients who screen positive for PTE will have an in-depth clinical visit
  Groups: Abbreviated Assessment Battery (AAB); Comprehensive Assessment Battery (CAB)
Procedure: Blood Draw — Blood Draw for Plasma, DNA, Serum, RNA
  Groups: Abbreviated Assessment Battery (AAB); Comprehensive Assessment Battery (CAB); TED Friend Controls
Procedure: EEG — An EEG will be performed on patients who screen positive for PTE at the clinical visit
  Groups: Abbreviated Assessment Battery (AAB); Comprehensive Assessment Battery (CAB)
Behavioral: Telephone Outcome Assessment — Assessments will be administered over the telephone to evaluate participant outcome status and screen for PTE
  Groups: Telephone Assessment Battery

SUMMARY:
The overarching goal of this study is to improve understanding of the long-range natural history of TBI and post-traumatic epilepsy (PTE) by extending follow-up of a previously enrolled cohort (TRACK-TBI) beyond the first 12 months after injury.

DETAILED DESCRIPTION:
This longitudinal observational study is part of the Transforming Research and Clinical Knowledge in Traumatic Brain Injury (TRACK-TBI) initiative, a multi-institutional project designed to characterize the acute and longer-term clinical, neuroimaging, and blood biomarker features of TBI. TRACK-TBI enrolled TBI patients at 18 Level 1 Trauma Centers in the US, across the age and injury spectrum. This study will extend the follow-up period for TRACK-TBI participants. The extensive clinical, imaging, and biomarker data that has already been collected in these TRACK-TBI participants, in combination with the extended longitudinal data, will allow for the identification of risk factors, co-morbidities, and prognostic biomarkers of TBI. Consequently, the extension of study follow-up will help to determine negative neurological and psychological outcomes of individuals who experienced a TBI compared to healthy and orthopedic controls.

The TRACK-EPI project aims to address the gaps in the existing literature and in the TRACK project regarding PTE. Post-traumatic epilepsy (PTE) is a common complication of traumatic brain injury (TBI), occurring in up to 20% of civilian patients and as many as 50% of military service members who suffer severe brain trauma, and 3-5% of those who suffer moderate TBI. Epilepsy resulting from brain trauma is often difficult to control with medical therapy, and is the cause of epilepsy in approximately 5% of patients referred to specialized epilepsy centers. PTE can be the result of TBI of any severity, although the risk is higher from severe TBI. PTE can arise through a variety of mechanisms, which may co-exist within a single patient. Focal brain injury, which results from penetrating trauma or focal contusions can result in epileptogenesis. Closed head injury can also produce diffuse injury, with shearing of axons and blood vessels, diffuse edema and ischemia, and secondary cellular damage through the release of inflammatory mediators. The clinical features of epilepsy, such as the frequency and severity of seizures, prevalence of associated co-morbidities, and responsiveness to therapy, may differ among these diverse mechanisms. Additionally, the neurophysiologic and imaging features of epileptogenicity also likely differ. Given the frequency of PTE, a more complete understanding of PTE etiology and prognosis is vital. Furthermore, it is likely that a sophisticated understanding of the subtypes of epilepsy resulting from brain trauma will be required to successfully develop anti-epileptogenic therapies.

ELIGIBILITY:
Inclusion Criteria:

Cohort TBI subjects with PTE

1. Participation in TRACK-TBI Observational Study (Penn IRB # 825503 or local IRB) and/or Spreading Depolarizations II (SDII) (Penn IRB # 828395 or local IRB) who are at least two years post-injury and completed at least 1 GOSE during the TRACK-TBI follow-up assessments
2. Must complete at least one Telephone Assessment (and a recruitment phone call)
3. Endorsed any one of four post-traumatic epilepsy (PTE) items from the Patient Interview at the 6 month or later TRACK-TBI follow-up assessment, and did not have a diagnosis of epilepsy prior to the index TBI
4. Ability of participant or legally authorized representative to provide informed consent Cohort Orthopedic Controls

1. Participation in TRACK-TBI Observational Study (Penn IRB # 825503 or local IRB) and/or Spreading Depolarizations II (SDII) (Penn IRB # 828395 or local IRB) who are at least two years post-injury and completed at least 1 GOSE during the TRACK-TBI follow-up assessments 2. Must complete at least one Telephone Assessment (and a recruitment phone call) 3. Endorsed any one of four post-traumatic epilepsy (PTE) items from the Patient Interview at the 6 month or later TRACK-TBI follow-up assessment, and did not have a diagnosis of epilepsy prior to the index TBI 4. Ability of participant or legally authorized representative to provide informed consent 5. Initial TRACK-TBI orthopedic injury Cohort Friend Controls

1. Participation in TRACK-TBI Observational Study (Penn IRB # 825503 or local IRB) who are at least two years post-enrollment and completed at least 1 MRI during the TRACK-TBI follow-up assessments
2. Ability of participant or legally authorized representative to provide informed consent Participation in TED: Friend Controls Study (IRB # 827537)

Exclusion Criteria:

1. Epilepsy diagnosed prior to index TBI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants enrolled in TRACK-TBI who screen positive for PTE or participants enrolled in TED Friend Controls cohort
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Glasgow Outcome Scale Extended (GOSE) | 4-6 years after TRACK-TBI enrollment
  The GOSE provides an overall measure of functional status based on information on cognition, independence, employability, and social/community participation collected via structured interview. Individuals are described by one of the eight outcome categories: Dead (1); Vegetative State (2); Lower Severe Disability (3); Upper Severe Disability (4); Lower Moderate Disability (5); Upper Moderate Disability (6); Lower Good Recovery (7) and Upper Good Recovery (8). Good Recovery is defined as a score of 7-8, Moderate Disability is defined by a score of 5-6 and Severe Disability is defined by a score of 3-4.
Diagnostic Interview for Seizure Classification Outside of Video EEG Recording (DISCOVER) | 4-6 years after TRACK-TBI enrollment
  During the clinical evaluation, participants and their caregivers are educated about the heterogeneous and protean manifestations of epileptic seizures, and encouraged to contact study staff if seizures or seizure-like events are noted. The DISCOVER form has been found to be highly accurate when compared to gold-standard video-EEG recording in an Epilepsy Monitoring Unit for classifying seizures

SECONDARY OUTCOMES:
Serum NF-L (neurofilament light chain) | 4-6 years after TRACK-TBI enrollment
  Using advanced blood-based assay platforms, levels of blood biomarkers neurofilament light chain (NF-L) will be measured to validate the utility as a biomarkers for traumatic axonal injury (TAI).

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of California, San Francisco, San Francisco, California
  - Spaulding Rehabilitation Hospital, Charlestown, Massachusetts
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pennsylvania/Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas at Austin, Austin, Texas
  - University of Texas Southwestern, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No